CLINICAL TRIAL: NCT00845429
Title: Immunogenicity of Two Dosages of a Split, Cell-Based, Inactivated, Trivalent Influenza Vaccine Administered in Healthy Adult Subjects Aged 18 to 49 Years
Brief Title: Immunogenicity of a Split, Cell-Based, Inactivated, Trivalent Influenza Vaccine in Healthy Adult Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: GCE03
Record Dates: First submitted 2009-02-13; First posted 2009-02-18 (Estimated); Results first posted 2012-12-17 (Estimated); Last update posted 2012-12-19 (Estimated); Status verified 2012-12

CONDITIONS: Influenza; Orthomyxoviruses; Myxovirus Infection
Keywords: Influenza; Orthomyxoviruses; Split-virion inactivated influenza vaccine; cell-based vaccine; Adults
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1: Standard-dose Cell-based Influenza Vaccine (Experimental): Participants will receive a single dose of standard-dose cell-based influenza virus vaccine.
  Interventions: Biological: Influenza virus vaccine - cell based (2007-2008 Formulation)
- Group 2: High-dose Cell-based Influenza Vaccine (Experimental): Participants will receive a single dose of high-dose cell-based influenza virus vaccine.
  Interventions: Biological: Influenza virus vaccine - cell-based (2007-2008 Formulation)
- Group 3: Licensed Fluzone® Influenza Vaccine (Active Comparator): Participants will receive a single dose of licensed Fluzone® influenza vaccine.
  Interventions: Biological: Influenza virus vaccine (2007-2008 Formulation)

INTERVENTIONS:
Biological: Influenza virus vaccine - cell based (2007-2008 Formulation) — 0.5 mL, Intramuscular
  Arms: Group 1: Standard-dose Cell-based Influenza Vaccine
Biological: Influenza virus vaccine - cell-based (2007-2008 Formulation) — 1.0 mL, Intramuscular
  Arms: Group 2: High-dose Cell-based Influenza Vaccine
Biological: Influenza virus vaccine (2007-2008 Formulation) — 0.5 mL, Intramuscular
  Other Names: Fluzone® (2007-2008 formulation)
  Arms: Group 3: Licensed Fluzone® Influenza Vaccine

SUMMARY:
Primary Objective:

To describe the immune response to a single administration of 2 formulations of the investigational cell-based influenza vaccines in healthy adult subjects.

Secondary Objective:

To describe the safety following a single administration of 2 formulations of the investigational cell-based influenza vaccines in healthy adult subjects.

DETAILED DESCRIPTION:
This is a multi-center study in healthy adult subjects. All subjects will receive a single dose of one of the influenza vaccine formulations and will provide blood samples for immunogenicity assessment.

ELIGIBILITY:
Inclusion Criteria :

* Healthy male or female subject, aged ≥ 18 to < 50 years on the day of inclusion
* Informed consent form signed
* Able to attend all scheduled visits and to comply with all trial procedures
* For a woman of childbearing potential: a negative urine pregnancy test and documented use of an effective method of contraception or abstinence for at least four weeks pre vaccination and up until three weeks post-vaccination

Exclusion Criteria :

* Subject currently breast-feeding.
* Participation in another clinical trial investigating a vaccine, drug, medical device, or medical procedure in the 4 weeks preceding the trial vaccination.
* Planned participation in another clinical trial during the present trial period.
* Prior participation in the Phase I trial of FLU INTERPAN (PER.C6) vaccine (study GCE01).
* Congenital or history of acquired immunodeficiency, or immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months.
* Systemic corticosteroid therapy as except the use of topical or inhalant corticosteroids
* Systemic hypersensitivity to egg proteins, chicken proteins, or to any of the vaccine components, or history of a life-threatening reaction to the trial vaccine or a vaccine containing the same substances.
* Chronic illness at a stage that could interfere with trial conduct or completion (chronic illness may include, but is not limited to, cardiac, renal or auto-immune disorders, or diabetes).
* Receipt of blood or blood-derived products in the 3 months preceding vaccination.
* Receipt of any vaccination in the 4 weeks preceding vaccination, or planned receipt of any vaccination in the 4 weeks following the trial vaccination.
* History of influenza infection (confirmed either clinically, serologically or microbiologically) within the 6 months preceding vaccination.
* Previous vaccination against influenza (in the 6 months preceding the trial vaccination).
* Planned receipt of any other 2007-2008 influenza vaccine.
* Thrombocytopenia or bleeding disorder contraindicating intramuscular (IM) vaccination.
* Subject deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized without his/her consent.
* History of Guillain-Barré syndrome
* Current abuse of alcohol or drug addiction that may interfere with the subject's ability to comply with trial procedures
* Any other condition which in the opinion of the investigator would pose a health risk to the participant or interfere with the evaluation of the vaccine.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 729 (Actual)
Dates: Start 2007-10; Primary Completion 2008-08 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (15):
- United States (15):
  - Hoover, Alabama
  - Mobile, Alabama
  - Tucson, Arizona
  - Milford, Connecticut
  - Pinellas Park, Florida
  - Chicago, Illinois
  - Wichita, Kansas
  - Kansas City, Missouri
  - Springfield, Missouri
  - Cary, North Carolina
  - Raleigh, North Carolina
  - Cincinnati, Ohio
  - Bensalem, Pennsylvania
  - Warwick, Rhode Island
  - Mt. Pleasant, South Carolina

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 16 to 23 October 2007 in 15 clinical centers in the US.
Pre-assignment Details: A total of 729 participants who met the inclusion, but no exclusion criteria were enrolled and vaccinated.
Groups:
- Group 1: Standard Dose Cell-Based Influenza Vaccine: Participants received a single dose of standard-dose cell-based influenza vaccine; 0.5 ml, intramuscularly.
- Group 2: High-dose Cell-Based Influenza Vaccine: Participants received a single dose of high-dose cell-based influenza vaccine; 1.0 ml, intramuscularly.
- Group 3: Licensed Fluzone® Influenza Vaccine: Participants received a single dose of licensed Fluzone® influenza vaccine; 0.5 ml, intramuscularly.
Period: Overall Study
Arm/Group | Group 1: Standard Dose Cell-Based Influenza Vaccine | Group 2: High-dose Cell-Based Influenza Vaccine | Group 3: Licensed Fluzone® Influenza Vaccine
Started | 244 | 241 | 244
Completed | 230 | 226 | 224
Not Completed | 14 | 15 | 20
Not completed — Protocol Violation | 5 | 4 | 7
Not completed — Lost to Follow-up | 7 | 9 | 10
Not completed — Withdrawal by Subject | 2 | 2 | 2
Not completed — Serious adverse event | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Standard Dose Cell-Based Influenza Vaccine | Group 2: High-dose Cell-Based Influenza Vaccine | Group 3: Licensed Fluzone® Influenza Vaccine | Total
Number analyzed (Participants) | 244 | 241 | 244 | 729
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 244 | 241 | 244 | 729
  >=65 years | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: Years] | 34.4 (9.41) | 34.5 (9.18) | 34.1 (9.42) | 34.3 (9.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 158 | 162 | 151 | 471
  Male | 86 | 79 | 93 | 258
Region of Enrollment [Number; unit: participants]
  United States | 244 | 241 | 244 | 729

OUTCOME MEASURES:

1. Primary Outcome: Summary of the Pre- and Post-Vaccination Geometric Mean Titers (GMTs) for Each of the Influenza Vaccine Antigens.
Time Frame: Days 0 and 21 post-vaccination
Population: Geometric mean titers were assessed in the full analysis set population.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Group 1: Standard Dose Cell-Based Influenza Vaccine | Group 2: High-dose Cell-Based Influenza Vaccine | Group 3: Licensed Fluzone® Influenza Vaccine
Number analyzed (Participants) | 236 | 233 | 238
Titers
  A/H1N1: Solomon Islands, Day 0 (N = 236, 231, 237) | 25.9 [21.0 to 32.0] | 26.4 [21.6 to 32.4] | 26.6 [21.7 to 32.5]
  A/H1N1: Solomon Islands, Day 21 (N= 236, 232, 238) | 184.8 [150.1 to 227.5] | 226.6 [187.2 to 274.4] | 425.1 [357.2 to 505.9]
  A/H3N2: Wisconsin, Day 0 (N = 236, 232, 237) | 51.2 [41.2 to 63.6] | 53.4 [43.8 to 65.2] | 51.5 [41.4 to 64.0]
  A/H3N2: Wisconsin, Day 21 (N = 236, 230, 238) | 288.3 [243.1 to 342.0] | 351.3 [302.2 to 408.5] | 692.4 [596.3 to 803.9]
  B: Malaysia, Day 0 (N = 236, 233, 238) | 13.4 [11.8 to 15.1] | 14.3 [12.6 to 16.3] | 14.2 [12.5 to 16.2]
  B: Malaysia, Day 21 (nN= 235, 233, 237) | 51.1 [43.2 to 60.4] | 53.0 [45.6 to 61.6] | 108.6 [95.4 to 123.7]

2. Primary Outcome: Percentage of Participants With Seroprotection to Each of the Influenza Vaccine Antigen Before and Post-vaccination.
Description: Seroprotection was defined as a titer ≥ 40 1/dil, and determined in participants with a valid serology result for the particular Flu strain, including results reported as less than lower limit of quantitation (LLOQ)
Time Frame: Day 21 post-vaccination
Population: Seroprotection was assessed in the full analysis set population.
Measure: Number; unit: Percentage of Participants
Arm/Group | Group 1: Standard Dose Cell-Based Influenza Vaccine | Group 2: High-dose Cell-Based Influenza Vaccine | Group 3: Licensed Fluzone® Influenza Vaccine
Number analyzed (Participants) | 236 | 233 | 238
Percentage of Participants
  A/H1N1: Solomon Islands Day 0 (N = 236, 231, 237) | 40 | 39 | 41
  A/H1N1: Solomon Islands Day 21 (N = 236, 232, 238) | 86 | 90 | 98
  A/H3N2: Wisconsin Day 0 (N = 236, 232, 237) | 54 | 62 | 55
  A/H3N2: Wisconsin Day 21 (N = 236, 230, 238) | 94 | 98 | 99
  B: Malaysia Day 0 (N = 236, 233, 238) | 14 | 20 | 20
  B: Malaysia Day 21 (N = 235, 233, 237) | 60 | 64 | 87

3. Primary Outcome: Percentage of Participants Achieving Seroconversion or Significant Increase at Day 21 Following Vaccination With Influenza Vaccine.
Description: Seroconversion: For participants with a Day 0 pre-vaccination titer < 10 (1/dil), titer ≥ 40 (1/dil) on Day 21.
  Significant Increase: For participants with a Day 0 pre-vaccination titer ≥ 10 (1/dil), ≥ 4-fold increase of titer on Day 21.
Time Frame: Day 21 post-vaccination
Population: Seroconversion and significant increase in Influenza vaccine antibodies were assessed in the full analysis set population.
Measure: Number; unit: Percentage of Participants
Arm/Group | Group 1: Standard Dose Cell-Based Influenza Vaccine | Group 2: High-dose Cell-Based Influenza Vaccine | Group 3: Licensed Fluzone® Influenza Vaccine
Number analyzed (Participants) | 236 | 233 | 238
Percentage of Participants
  A/H1N1: Solomon Islands (N = 236, 231, 237) | 54 | 63 | 74
  A/H3N2: Wisconsin (N = 236, 230, 237) | 50 | 53 | 71
  B: Malaysia (N = 235, 233, 237) | 38 | 38 | 61

4. Secondary Outcome: Number of Participants Reporting at Least 1 Solicited Injection Site or Systemic Reaction Post-vaccination With Influenza Vaccine.
Description: Solicited Injection Site Reactions: Pain, erythema or redness, swelling, ecchymosis, and induration.
  Solicited Systemic Reactions: Fever (temperature), headache, malaise, myalgia, and rigors.
Time Frame: Day 0 up to Day 7 post-vaccination
Population: Safety analysis was on all enrolled and vaccinated participants with available reaction data, intent-to-treat population.
Measure: Number; unit: Participants
Arm/Group | Group 1: Standard Dose Cell-Based Influenza Vaccine | Group 2: High-dose Cell-Based Influenza Vaccine | Group 3: Licensed Fluzone® Influenza Vaccine
Number analyzed (Participants) | 244 | 241 | 244
Participants
  Any Solicited Injection Site Reaction | 117 | 156 | 184
  Any Pain | 103 | 144 | 175
  Grade 3 Pain (incapacitating, prevents activities) | 1 | 2 | 1
  Any Erythema | 36 | 57 | 55
  Grade 3 Erythema (≥ 5 cm) | 0 | 0 | 4
  Any Swelling | 24 | 23 | 36
  Grade 3 Swelling (≥ 5 cm) | 0 | 0 | 1
  Any Ecchymosis | 6 | 19 | 14
  Grade 3 Ecchymosis (≥ 5 cm) | 0 | 0 | 1
  Any Induration | 31 | 29 | 38
  Grade 3 Induration (≥ 5 cm) | 0 | 0 | 0
  Any Solicited Systemic Reaction | 114 | 126 | 137
  Any Fever | 13 | 9 | 11
  Grade 3 Fever (39.0 ºC or 102.2 ºF) | 0 | 0 | 2
  Any Headache | 75 | 85 | 89
  Grade 3 Headache (Prevents daily activities) | 3 | 3 | 6
  Any Malaise | 58 | 54 | 63
  Grade 3 Malaise (Prevents daily activities) | 6 | 4 | 5
  Any Myalgia | 60 | 70 | 83
  Grade 3 Myalgia (Prevents daily activities) | 1 | 3 | 4
  Any Rigors | 16 | 9 | 13
  Grade 3 Rigors (Prevents daily activities) | 2 | 1 | 1

ADVERSE EVENTS:
Time Frame: Adverse events data were collected from the day of vaccination (Day 0) to up to 6 months post-vaccination.
Arm/Group | Group 1: Standard Dose Cell-Based Influenza Vaccine | Group 2: High-dose Cell-Based Influenza Vaccine | Group 3: Licensed Fluzone® Influenza Vaccine
Serious Adverse Events (participants affected / at risk) | 3/244 | 4/241 | 6/244
Other Adverse Events (participants affected / at risk) | 158/244 | 179/241 | 199/244
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Standard Dose Cell-Based Influenza Vaccine (N=244) | Group 2: High-dose Cell-Based Influenza Vaccine (N=241) | Group 3: Licensed Fluzone® Influenza Vaccine (N=244)
Biliary Dyskinesia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Gallbladder Non-functioning (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Gastrointestinal Stoma Complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Pelvic Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Tibia Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Loss of Consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Ovarian Cyst Ruptured (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Group 1: Standard Dose Cell-Based Influenza Vaccine (N=244) | Group 2: High-dose Cell-Based Influenza Vaccine (N=241) | Group 3: Licensed Fluzone® Influenza Vaccine (N=244)
Injection site Pain (General disorders) | 103/240 | 144/234 | 175/238
Injection site Erythema (General disorders) | 36/240 | 57/234 | 55/238
Injection site Swelling (General disorders) | 24/240 | 23/234 | 36/238
Injection site Ecchymosis (General disorders) | 6/240 | 19/234 | 14/238
Injection site Induration (General disorders) | 31/240 | 29/234 | 38/238
Fever (General disorders) | 13/240 | 9/234 | 11/238
Malaise (General disorders) | 58/240 | 54/234 | 63/238
Rigors (General disorders) | 16/240 | 9/234 | 13/238
Myalgia (Musculoskeletal and connective tissue disorders) | 60/240 | 70/234 | 83/238
Headache (Nervous system disorders) | 75/240 | 85/234 | 89/238

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.